CLINICAL TRIAL: NCT02181959
Title: Safety and Tolerability of PHARMATON Capsules vs PHARMATON Capsules With DMAE vs Placebo in Healthy Volunteers (A Double-blind, Controlled Multicentre Study)
Brief Title: Safety and Tolerability of Pharmaton Capsules in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1114.10
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- Pharmaton® with DMAE (Experimental)
  Interventions: Drug: Pharmaton® with DMAE
- Pharmaton® without DMAE (Active Comparator)
  Interventions: Drug: Pharmaton® without DMAE
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pharmaton® with DMAE
  Arms: Pharmaton® with DMAE
Drug: Pharmaton® without DMAE
  Arms: Pharmaton® without DMAE
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this trial was to evaluate the safety and tolerability of a galenic formulation of Pharmaton® capsules containing 2-Dimethylaminoethanol (DMAE) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman, between 20 to 70 years
* Fit to work
* Volunteers have given informed consent and signed the consent form

Exclusion Criteria:

* Any serious disorder that might interfere with his/her participation in this study and the evaluation of the safety of the test drug (e.g. renal insufficiency, hepatic dysfunction, cardiovascular disease, disorders of the calcium metabolism, hypervitaminosis A or D, psychic disorder, etc)
* Treatment with other drugs that might interfere with the evaluation of the safety of the test drug
* Known hypersensitivity to any ingredients of the study drug
* Pregnancy, lactation, women of childbearing potential who do not use an established contraceptive
* Drug and alcohol abuse
* Participation in another trial
* Known abnormal values of the laboratory tests (if detected after enrolment, subjects will continue the treatment provided there are no medical objections)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 1998-12; Primary Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 60 days
Assessment of overall tolerability rate on a 4-point scale | Day 30 and 60

SECONDARY OUTCOMES:
Number of patients with abnormal changes in laboratory parameters | Day 0, 30 and 60
Number of patients with abnormal findings in physical examination | Day 0, 30 and 60